CLINICAL TRIAL: NCT01997424
Title: Association of Non-alcoholic Fatty Liver Disease and Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Principal Investigator, Georg Dultz, MD, Johann Wolfgang Goethe University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: JWGUHMED1-007
Record Dates: First submitted 2013-10-23; First posted 2013-11-28 (Estimated); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Non-alcoholic Fatty Liver Disease (NAFLD)
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Controlled Attenuation Parameter (CAP), Echosens, Paris, France
Device: FibroScan, Echosens, Paris, France

SUMMARY:
This study will evaluate the association of non-alcoholic fatty liver disease and diabetes mellitus. Patients presenting in our clinic with Diabetes mellitus type 1 or 2 will receive the following examination:

* Transient Elastography and Controlled Attenuation Parameter using the FibroScan
* blood examination including biochemical markers The statistically calculated sample size needed is 340 patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 years and older
* Written informed consent
* Diabetes mellitus type 1 or 2

Exclusion Criteria:

* Patients with mental diseases
* Pregnancy or lactation
* Ascites
* Continued alcohol consumption (> 21 drinks/week for male and > 14 drinks/week for female patients)
* Chronic liver disease (viral hepatitis, autoimmune hepatitis, PBC, PSC, hemochromatosis, M Wilson)
* Hepatocellular carcinoma/ Liver metastasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Actual)
Dates: Start 2013-05; Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Steatosis | one day
  • Evaluating the presence of liver steatosis in patients with diabetes mellitus using the ultrasound-based method "Controlled Attenuation Parameter", which is integrated in the FibroScan machine and can non-invasively quantify liver steatosis (Steatosis fibrosis scores I-III [ Designated as safety issue: No ]; Steatosis scores: 0 = <5% I = 5-33% II = 33-66% III = >66%)

SECONDARY OUTCOMES:
Fibrosis | one day
  • Evaluation of the prevalence of liver fibrosis using transientelastography (FibroScan) and serological markers in patients with diabetes mellitus (Liver fibrosis scores I-IV (METAVIR) [ Designated as safety issue: No ]; METAVIR fibrosis scores: I = mild fibrosis II = significant fibrosis III = advanced fibrosis IV = cirrhosis)
Steatosis (serum) | one day
  • Evaluating the prevalence of liver steatosis using serum steatosis markers in patients with diabetes mellitus

CONTACTS AND LOCATIONS:
Overall Officials: Mireen Friedrich-Rust, MD, Principal Investigator — Goethe University
Locations (1):
- University Hospital Frankfurt, Frankfurt am Main, Hesse, Germany